CLINICAL TRIAL: NCT04683991
Title: The Effect of Different Surgical Timing on the Clinical Efficacy of Increasing the Thickness of Keratinized Mucosa Around a Single Posterior Implant: a Prospective, Randomized Controlled Clinical Trial
Brief Title: Increased Peri-implant Keratinized Mucosal Thickness at Different Operative Times
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-782
Record Dates: First submitted 2020-12-22; First posted 2020-12-24 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-01

CONDITIONS: Dental Implants; Peri-Implantitis
Keywords: keratinized mucosa thickness; dental Implants; subepithelial connective tissue graft; marginal bone level
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: 1:1 randomized controlled clinical trial were used. Random numbers generated by SPSS26.0 will be placed in sequentially coded, sealed, opaque envelopes. Only "1" or "0" will be generated, and the number of "1" or "0" generated by SPSS26.0 is 17. When the qualifications of the subjects were determined by the researchers, the envelopes were opened sequentially and the subjects were assigned to groups. The number "1" represented the treatment group 1 and the number "0" represented the treatment group 2.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group 1 (Experimental): At the same time of implant implantation, autologous tissue is transplanted into the recipient area by using Subepithelial connective tissue graft.
  Interventions: Procedure: Subepithelial connective tissue graft
- treatment group 2 (Experimental): During the second stage operation, autologous tissue is transplanted into the recipient area by using Subepithelial connective tissue graft.
  Interventions: Procedure: Subepithelial connective tissue graft

INTERVENTIONS:
Procedure: Subepithelial connective tissue graft — A de-epithelialized connective tissue graft is harvested from the homolateral palate and transplanted around the implant.

SUMMARY:
Keratinized mucosa, which is composed of free gingiva and attached gingiva, is a barrier against bacterial invasion in oral cavity and provides good tissue sealing for periodontal environment. When the keratinized mucosa is insufficient, it is difficult to maintain the long-term stability of the implant, which is not conducive to the peri-implant health. It is generally believed that enough keratinized mucosa width is beneficial to reduce plaque accumulation and reduce the incidence rate of peri-implant diseases. In recent years, clinicians have gradually recognized that the thickness of keratinized mucosa plays an important role in maintaining the peri-implant health. Some researchers found that the thickness of mucosa is very important to maintain the aesthetic effect of implant restoration, and when the thickness of mucosa around the implant is less than 2mm, alveolar bone absorption will occur to maintain a stable biological width. A meta-analysis showed that when the thickness of the keratinized mucosa around the implant was greater than 2mm, the amount of marginal bone loss was significantly reduced (- 0.8mm, P < 0.0001).

It is considered that autogenous soft tissue graft is the most reliable technology to augment keratinized mucosa. Subepithelial connective tissue graft (SCTG) is a mucogingival surgery that transplant autologous free connective tissue under the pedicled semi thick flap to augment keratinized mucosa. It can effectively increase the thickness of soft tissue, cover the exposed implant, and reconstruct the interdental papilla. It is the gold standard for peri-implant soft tissue agumentation. Keratinized mucosal thickening surgery may be done prior to the surgical phase, after the surgical phase, before loading, or even after loading. It is believed that keratinized mucosal thickening at the same time of implantation can effectively reduce the possibility of mucosal recession after implantation, reduce the amount of marginal bone absorption in the process of osseointegration, which is conducive to maintaining the long-term stability of the implant. For the sake of clear clinical vision and convenient operation, clinicians often choose to thicken the keratinized mucosa during the secondary operation, and also obtain good postoperative effect. However, after the completion of the final repair, the keratinized mucosa thickening surgery increases the difficulty of operation and the technical requirements for the operator. In clinical practice, it is rarely selected to perform keratinized mucosal thickening at this time. At present, the effectiveness of timing on the outcome of soft tissue augmentation is still debated, and, most importantly, a direct comparison between simultaneous and staged procedures remains underexplored.

Therefore, this clinical trial is to prospectively compare the clinical efficacy of simultaneous versus delayed timing of soft tissue augmentation by SCTG placement around single implants, by evaluating the peri-implant marginal bone level change and soft tissue change, so as to provide reference for the formulation of clinical treatment plan and the selection of the best operation time.

ELIGIBILITY:
Inclusion Criteria:

* No systemic diseases or pregnancy;
* The thickness of keratinized mucosa where the posterior tooth is missing is less than 2 mm;
* Full-mouth plaque score (FMPS) < 20% (measured at four sites per tooth) and bleeding on probing score (BOP%) ≤25% (measured at six sites per tooth);
* Periodontal condition is stable, no probing depths ≥5 mm;
* No previous soft tissue augmentation procedure at experimental site;
* The patient has signed informed consent and accepts the operation of subepithelial connective tissue transplantation.

Exclusion Criteria:

* Patients with uncontrolled hypertension;
* Patients with uncontrolled diabetes;
* Patients with insufficient oral hygiene and Untreated periodontitis;
* Pregnant or lactating women;
* Smoker;
* Patients with long-term (> 6 months) use of glucocorticoids;
* History of malignancy, radiotherapy, or chemotherapy for malignancy within the past 5 years;
* Patients with severe cardiovascular problems;
* Patients with uncontrolled infectious or metabolic diseases;
* Patients with substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
peri-implant marginal bone level change | 18 months
  The bone level of the proximal and distal sites of the implant is measured by oral X-ray parallel projection method. Compare the image value with the actual value to calculate the actual bone level.

SECONDARY OUTCOMES:
peri-implant clinical attachment level change | 18 months
  The distance between the reference point of impression edge and the bottom of gingival groove around the implant.
peri-implant keratinized mucosa width | 18 months
  keratinized tissue measured as the distance between muco-gingival junction and the gingival margin.
peri-implant keratinized mucosa thickness | 18 months
  gingival thickness measured 1.5 mm coronal to the MGJ using an injection needle, perpendicular to the tissue surface, with a silicon stop over the gingival surface.
peri-implant gingival index | 18 months
  Periodontal probe was used to measure 6 sites on buccal and lingual side each time to observe gingival color, texture and bleeding, and record the scores.
peri-implant gingival recession | 18 months
  The distance between the implant shoulder and the gingival margin of the temporary or final crown was measured with a periodontal probe (only when the implant shoulder was visible).
visual analogue scale | 18 months
  Visual analogous scale ( VAS) suggested by WHO was used to assess. Analgesia intensity expressed with 0-10, 0 point as without pain completely, 10 points as unbearable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Weilian Sun, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Department of Oral Medicine, the Second Affiliated Hospital, School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No